CLINICAL TRIAL: NCT00503659
Title: Comparison of Two Methods of Bronchial Methacholine Provocation: PC 20 FEV1 Versus PD 20 FEV1
Brief Title: Comparison of Two Methods of Bronchial Methacholine Provocation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johann Wolfgang Goethe University Hospital (Other)
Responsible Party: Principal Investigator, Johannes Schulze MD, Consultant Pediatric Allergy and Pulmonológy, Johann Wolfgang Goethe University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 335/06/FFM
Record Dates: First submitted 2007-07-18; First posted 2007-07-19 (Estimated); Last update posted 2011-10-12 (Estimated); Status verified 2011-10

CONDITIONS: Bronchial Hyperreactivity; Bronchial Asthma
Keywords: PC20 FEV1; PD20FEV1; bronchial hyperreactivity; bronchial asthma
MeSH Terms: conditions — Bronchial Hyperreactivity; Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Active Comparator): Methacholine challenge, five-breath dosimeter protocol
  Interventions: Procedure: Bronchial methacholine provocation
- B (Active Comparator): Methacholine challenge five incremental dosages protocol
  Interventions: Procedure: Bronchial methacholine provocation

INTERVENTIONS:
Procedure: Bronchial methacholine provocation — A short five-breath dosimeter protocol using a five-step dilution schedule according to ATS guidelines (0.0625, 0.25, 1, 4, 16 mg/ml methacholine)
  Other Names: DeVilbiss nebulizer
  Arms: A
Procedure: Bronchial methacholine provocation — A five-step protocol using a single dilution of 16 mg/ml methacholine (0.01, 0.1, 0.4, 0.8, 1.6 mg)
  Other Names: Viasys APS nebulizer
  Arms: B

SUMMARY:
This study is meant to compare two routine diagnostic approaches in patients with bronchial asthma. Patients are challenged with methacholine in order to measure their bronchial response. We compare the evaluation of the effects of incremental concentrations versus incremental dosages.

DETAILED DESCRIPTION:
Bronchial methacholine challenge is well established in asthma diagnostic and research purposes. ATS guidelines provide a short five-breath dosimeter protocol using a five-step dilution schedule. The Viasys APS system enables a feasible and less time consuming provocation with incremental dosages. In 48 young adults with bronchial hyperreactivity (BHR) the ATS-protocol with a five-step protocol using a single dilution of 16 mg/ml methacholine should be compared.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent
* Age 12-45 years
* Known bronchial hyperreactivity

Exclusion Criteria:

* Age < 12 > 45 years
* Clinical asthma requiring regular inhalation
* Vital capacity < 80%
* FEV1 < 75%
* Chronic disease conditions or infections
* Pregnancy
* Inhalative or systemic steroid use
* Substance abuse
* Incapability of understanding the study's purpose and performance

Ages: 12 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 48 (Actual)
Dates: Start 2007-02; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
correlation of the two parameters PC20 FEV1 and PD20 FEV1 | feb 2007 - dec 2007

SECONDARY OUTCOMES:
kappa index of concordance: reliability of the two procedures as to a FEV1 decrease of 20% depending on methacholine concentration | see above

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Zielen, M.D., Ph.D., Principal Investigator — Goethe University, Department of Pulmonology
Locations (1):
- Goethe University, Department of Pulmonology, Frankfurt am Main, Hesse, Germany

REFERENCES:
- [Background] Crapo RO, Casaburi R, Coates AL, Enright PL, Hankinson JL, Irvin CG, MacIntyre NR, McKay RT, Wanger JS, Anderson SD, Cockcroft DW, Fish JE, Sterk PJ. Guidelines for methacholine and exercise challenge testing-1999. This official statement of the American Thoracic Society was adopted by the ATS Board of Directors, July 1999. Am J Respir Crit Care Med. 2000 Jan;161(1):309-29. doi: 10.1164/ajrccm.161.1.ats11-99. No abstract available. PMID 10619836